CLINICAL TRIAL: NCT04571008
Title: Effect of Nicotinamide Mononucleotide (NMN) Supplementation on Organ System Biology
Brief Title: Effect of NMN Supplementation on Organ System Biology
Acronym: VAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 201909118
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): At least 16 weeks of placebo.
  Interventions: Other: Placebo
- NMN supplementation (Experimental): At least 16 weeks of NMN.
  Interventions: Dietary Supplement: Treatment

INTERVENTIONS:
Other: Placebo — Intervention will last at least 16 weeks in the form of two capsules.
  Arms: Placebo
Dietary Supplement: Treatment — Intervention will last at least 16 weeks in the form of two or three NMN capsules (total of 300 or 450 mg/day).
  Arms: NMN supplementation

SUMMARY:
The goal of this proposal is to determine whether the beneficial effects of NMN on metabolic function observed in rodents applies to people.

DETAILED DESCRIPTION:
This study is looking at the effect of the dietary supplement "Nicotinamide mononucleotide" (NMN) on key cardiovascular and metabolic functions, specifically those that are important risk factors for diabetes and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25.0-50.0 kg/m²
* Prediabetes defined as fasting plasma glucose of ≥100 mg/dL, or HbA1C ≥5.7, or HOMA-IR ≥2.5.

Exclusion Criteria:

* Women who are still having menses
* Persons who take niacin, nicotinamide, or other vitamin B3-related supplementation and are not willing to discontinue supplementation for 3 weeks before medical screening and during the entire study period
* Persons who consume moderate-large amounts of caffeine daily (>2 cups of coffee or 8 oz caffeinated drinks per day) or consume less amounts of caffeine but believe withdrawal symptoms (e.g. headache) are likely if caffeine is stopped
* Unstable weight (>3% change during the last 2 months before entering the study)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Change in Muscle insulin sensitivity | before and after at least 16 weeks of treatment
  The outcome will be assessed during hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotopic tracer infusion before and after intervention period.

SECONDARY OUTCOMES:
Changes in glucose tolerance | before and after at least 16 weeks of treatment
  The outcome will be assessed during modified oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States